CLINICAL TRIAL: NCT02509975
Title: An Open Label, Single Center, Pilot Study to Evaluate the Safety and Effectiveness of OCL 503 in Prostate Artery Embolization for the Treatment of Men With Benign Prostatic Hypertrophy
Brief Title: Safety and Efficacy of OCL 503 in Prostate Artery Embolization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMBiotechnologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCL503-P2-PAE-01
Record Dates: First submitted 2015-07-24; First posted 2015-07-28 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Benign Prostatic Hyperplasia; Benign Prostatic Hypertrophy
Keywords: embolization; prostate
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prostate Artery Embolization (Experimental): Transarterial administration of OCL 503 to the arteries feeding the prostate.
  Interventions: Device: Prostate artery embolization.

INTERVENTIONS:
Device: Prostate artery embolization. — Embolization of the prostatic vasculature with OCL 503 using a microcatheter.

SUMMARY:
This is a prospective, pilot, open-label, uncontrolled, non-randomized safety and effectiveness study of OCL 503 in men with BPH.

DETAILED DESCRIPTION:
Prior to entering the study, all patients will undergo pre-study assessments including compliance with inclusion and exclusion criteria, laboratory assessments, IPSS, uroflowmetry, IIEF, and MRI pelvic imaging. Following conventional catheter angiography with cone-beam CT to confirm catheter placement and prostatic vasculature, each patient will undergo transarterial embolization with OCL 503. OCL 503 will be administered intra-arterially via microcatheter until there is stasis of blood flow.

Patient assessments include blood work, IPSS, uroflowmetry, IIEF, MRI and patient interviews conducted at 3 months, 6 months, and 12 months post embolization.

ELIGIBILITY:
Inclusion Criteria:

* Patient has received a diagnosis of BPH with moderate to severe LUTS, as determined by IPSS
* Patient is greater than 50 years of age
* Patient has had a pelvic examination within the past 6 months
* Patient has been refractory to medical therapy for the last 6 months, or has refused medical therapy
* Patient has a Qmax below 15 mL/s or acute urinary retention
* Prostate is larger than 40 cubic centimetres
* Patient is willing and able to provide written, informed consent

Exclusion Criteria:

* Known malignancy
* Serum PSA > 10 ng/mL at screening
* Advanced atherosclerosis and tortuosity of the iliac arteries
* Prior transurethral resection of the prostate (TURP)
* Post void retention (PVR) > 250 mL
* Chronic use of metronidizole
* Phytotherapy for BPH within last two weeks of screening visit
* Secondary renal insufficiency due to prostatic obstruction
* Chronic renal failure (GSR < 60)
* Large bladder diverticula or bladder stones
* Claustrophobia or other contraindications related to performing MRI
* Compromised hematopoietic function
* Anaphylactic reaction to drug or anesthetic, allergic reaction to iodine or contrast media
* Investigational drug or experimental therapy in the past 4 weeks
* Abnormal coagulation profile
* Allergy to bovine collagen

Min Age: 51 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Safety of OCL 503 as measured by Adverse Events reporting. | 12 months
  Measurement of device related adverse events post embolization of the prostatic vasculature, at 30 days.
International Prostate Symptom Score (IPSS) | 12 months
  Measurement of IPSS at 12 months post embolization of the prostatic vasculature with OCL 503.

SECONDARY OUTCOMES:
Tissue Response | 12 months
  Measurement in the change in size of the prostate by MRI at 12 months post embolization of the prostatic vasculature with OCL 503.
Uroflowmetry | 12 months
  Measurement of Qmax, post-voiding bladder retention (PVR) at 12 months post embolization of the prostatic vasculature with OCL 503.
International Index of Erectile Function (IIEF) | 12 months
  Measurement of IIEF by questionnaire at 12 months post embolization of the prostatic vasculature using OCL 503.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Owen, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada